CLINICAL TRIAL: NCT06457958
Title: The Effect of Sevoflurane and Desflurane Anesthetic Agents Used in Elective Cholecystectomy Surgery on Heme Oxygenase-1 mRNA Expression and Heme Oxygenase-1 Protein Levels: A Comparative Prospective Study
Brief Title: Effect of Sevoflurane and Desflurane on Heme Oxygenase-1 Expression in Elective Cholecystectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to lack of financial support.
Sponsor: Kocaeli City Hospital (Other Government)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KSH-ANREA-BG-01
Record Dates: First submitted 2024-06-01; First posted 2024-06-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Cholecystitis, Chronic
Keywords: Anesthetics, Inhalation; Heme Oxygenase-1; Oxidative Stress; Sevoflurane; Desflurane; Anesthesia, General; Cholecystectomy
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: There will be 2 parallel study arms where sevoflurane and desflurane are administered.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane Group (Active Comparator): Patients in this group will receive sevoflurane as the anesthetic agent during elective cholecystectomy surgery.
  Sevoflurane is a commonly used inhalational anesthetic known for its rapid onset and recovery times.
  Interventions: Drug: Sevoflurane Group
- Desflurane Group (Active Comparator): Patients in this group will receive desflurane as the anesthetic agent during elective cholecystectomy surgery.
  Desflurane is another widely used inhalational anesthetic, notable for its low blood-gas solubility coefficient, leading to very rapid onset and recovery times.
  Interventions: Drug: Desflurane Group

INTERVENTIONS:
Drug: Sevoflurane Group — Preoperative: One hour before surgery, a blood sample will be taken. Intraoperative: Sevoflurane will be used as the inhalational anesthetic. Routine general anesthesia procedures will be followed. Sevoflurane consumption, oxygen levels, and vital parameters will be recorded.
  Postoperative: One hour after extubation, another blood sample will be taken, marking the end of patient monitoring.
  Laboratory Analysis: Blood samples will be stored in the biochemistry laboratory. Hemoxygenase-1 protein levels will be measured by ELISA, and mRNA expression will be analyzed using PCR.
  Other Names: Sevoflurane maintenance anesthesia group
  Arms: Sevoflurane Group
Drug: Desflurane Group — Preoperative: One hour before surgery, a blood sample will be taken. Intraoperative: Desflurane will be used as the inhalational anesthetic. Routine general anesthesia procedures will be followed. Desflurane consumption, oxygen levels, and vital parameters will be recorded.
  Postoperative: One hour after extubation, another blood sample will be taken, marking the end of patient monitoring.
  Laboratory Analysis: Blood samples will be stored in the biochemistry laboratory. Hemoxygenase-1 protein levels will be measured by ELISA, and mRNA expression will be analyzed using PCR.
  Other Names: Desflurane maintenance anesthesia group
  Arms: Desflurane Group

SUMMARY:
General anesthesia is routinely administered to patients who undergo elective cholecystectomy. The most commonly used inhalation agents during general anesthesia are sevoflurane and desflurane. Participants who will undergo elective cholecystectomy surgery and meet the eligibility criteria will be randomized. Participants will be divided into two groups. One group will receive sevoflurane, and the other group will receive desflurane. Preoperative and postoperative blood samples will be taken from the participants. After the sample collection process is completed, the ELISA method will be used for measuring blood heme oxygenase-1 protein levels, and the PCR technique will be used for measuring blood heme oxygenase-1 mRNA gene expression. The increase in amounts between the two groups will be compared. This study aims to demonstrate the effects of the most commonly used inhalation agents on the levels of heme oxygenase-1 enzyme, which has been shown to be an important enzyme in cellular protection mechanisms, as well as on mRNA gene expression, and to determine which agent may be more effective in preventing cellular damage at the molecular level.

DETAILED DESCRIPTION:
In this study, the aim is to compare the effects of two commonly used inhalation agents, sevoflurane and desflurane, on heme oxygenase-1 (HO-1) enzyme levels. The total amounts of sevoflurane and desflurane administered to patients, as well as their overall oxygen consumption, will also be monitored. This data will allow for the exploration of how these inhalation agents and oxygen intake influence HO-1 enzyme levels, both across and within groups. The goal is to determine which agent demonstrates more effective cellular protection at the molecular level. This study will scientifically investigate how these commonly used agents impact HO-1 enzyme levels and gene expression, drawing conclusions based on the data obtained. The findings are anticipated to provide valuable insights for future clinical research and expand horizons in this field.

Study Design and Power Analysis:

The study follows a comparative prospective parallel-group design and is classified as low-risk scientific research. Sample size determination was based on a power analysis using G*Power 3.1 software. A t-test will be employed for comparison between two independent groups, with an alpha error probability set at 0.05 and a power (1-beta error probability) of 0.90. A total of 48 patients, with 24 in each group, will be included.

Inclusion Criteria:

Willing participants ASA class 1-2-3 Ages 18-65 Patients undergoing elective cholecystectomy surgery

Exclusion Criteria:

Patients undergoing emergency cholecystectomy surgery Pregnant and postpartum patients Patients with a history of oncological diseases Patients with known genetic diseases Patients receiving total intravenous anesthesia Patients developing complications during surgery

Study Procedures:

Preoperative blood samples will be obtained from enrolled patients 1 hour before surgery. Patients undergoing general anesthesia will be randomly assigned to receive either sevoflurane or desflurane inhalation agent. Standard anesthesia procedures will be followed. Total amounts of sevoflurane/desflurane consumed, oxygen consumption, and vital parameters will be recorded throughout the procedure. Postoperative blood samples will be collected 1 hour after extubation. Patient follow-up will then conclude. Blood samples will be stored in the hospital's biochemistry laboratory. HO-1 blood protein levels will be measured using the ELISA method, and HO-1 mRNA expression will be assessed using PCR. This study aims to determine which inhalation agent offers superior cellular protection at the molecular level by assessing their effects on HO-1 enzyme levels and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Willing participants
* ASA class 1-2-3
* Ages 18-65 years
* Patients undergoing elective cholecystectomy surgery

Exclusion Criteria:

* Patients undergoing emergency cholecystectomy surgery
* Pregnant and postpartum patients
* Patients with a history of oncological diseases
* Patients with known genetic diseases
* Patients receiving total intravenous anesthesia
* Patients developing complications during surgery will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Effects of Sevoflurane and Desflurane Inhalation Anesthetics on Blood Heme Oxygenase-1 Gene and Protein Levels | Postoperative at hour 1
  The aim of this study is to compare the effects of sevoflurane and desflurane, commonly used inhalation anesthetics in routine anesthesia practice, on blood heme oxygenase-1 gene and protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: BEDİRHAN GÜNEL, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, IZMIT, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request can be made to obtain patient data from the institution. Data will not be shared by the researchers.

REFERENCES:
- [Background] Bauer I, Raupach A. The Role of Heme Oxygenase-1 in Remote Ischemic and Anesthetic Organ Conditioning. Antioxidants (Basel). 2019 Sep 16;8(9):403. doi: 10.3390/antiox8090403. PMID 31527528
- [Background] Wu ZF, Lin WL, Lee MS, Hung NK, Huang YS, Chen TW, Lu CH. Propofol vs desflurane on the cytokine, matrix metalloproteinase-9, and heme oxygenase-1 response during living donor liver transplantation: A pilot study. Medicine (Baltimore). 2019 Nov;98(48):e18244. doi: 10.1097/MD.0000000000018244. PMID 31770287
- [Background] Hoetzel A, Schmidt R. Regulatory role of anesthetics on heme oxygenase-1. Curr Drug Targets. 2010 Dec;11(12):1495-503. doi: 10.2174/1389450111009011495. PMID 20704551